CLINICAL TRIAL: NCT06031012
Title: Compound Glutamine Enteric-Coated Capsules Combined with Thalidomide in Preventing Radiation-induced Oral Mucositis in Patients Undergoing Radiotherapy-a Multicenter, Open-label, Randomized Controlled Study
Brief Title: Compound Glutamine Enteric-Coated Capsules Combined with Thalidomide in Preventing Radiation-induced Oral Mucositis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Mei Shi, clinical professor of department of radiation oncology of XiJing hospital, Air Force Military Medical University, China
Allocation: Not Applicable | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AFMMUChina-oral mucocitis
Record Dates: First submitted 2023-08-29; First posted 2023-09-11 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Mucositis Oral
MeSH Terms: conditions — Stomatitis | interventions — Thalidomide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CGECC combined with thalidomide (Experimental): CGECC: Start oral administration on the first day of radiation therapy, continuing until one week after radiation therapy ends. Take three times a day, two tablets each time; once in the morning, once in the afternoon, and once in the evening.
  Thalidomide: Start oral administration on the first day of radiation therapy, continuing until one week after radiation therapy ends. Take orally at 100mg, once every evening.
  Interventions: Drug: CGECC combined with thalidomide
- CGECC alone (Active Comparator): CGECC: Start oral administration on the first day of radiation therapy, continuing until one week after radiation therapy ends. Take three times a day, two tablets each time; once in the morning, once in the afternoon, and once in the evening.
  Interventions: Drug: CGECC alone

INTERVENTIONS:
Drug: CGECC combined with thalidomide — Patients received glutamine combined with thalidomide from the beginning of radiotherapy to one week after radiotherapy.
  Other Names: GT group
  Arms: CGECC combined with thalidomide
Drug: CGECC alone — Patients received CGECC alone from the beginning of radiotherapy to one week after radiotherapy.
  Other Names: Cgroup
  Arms: CGECC alone

SUMMARY:
The goal of this study is to compare Compound Glutamine Enteric-Coated Capsules (CGECC) combined with thalidomide with CGECC in preventing radiation-induced oral mucositis. The aim of this study is to answer whether CGECC plus thalidomide could improve the median incidence time of grade 2 oral mucositis. Participants would be randomly divided into the two groups above mentioned.

DETAILED DESCRIPTION:
Explore the therapeutic efficacy of CGECC combined with Thalidomide as compared to CGECC alone in preventing radiation-induced oral mucositis. The primary research endpoint is the median time to the onset of Grade II oral mucositis, defined as the number of days from the start of radiation therapy to the occurrence of Grade II oral mucositis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years old;
2. Patients with postoperative oral malignant tumors confirmed by pathological histology or cytology and requiring radiotherapy;
3. Patients who have received more than 45Gy of radiation in the oral area;
4. ECOG PS (Eastern Cooperative Oncology Group Performance Status) score of 0-1;
5. Basic hematological indicators are normal: White blood cell count ≥ 4×10^9/L; Absolute neutrophil count ≥ 1.5×10^9/L; Platelets ≥ 100×10^9/L; Hemoglobin ≥ 90 g/L;
6. Basic renal function is normal: Serum creatinine ≤ 1.5×ULN (Upper Limit of Normal) or Creatinine Clearance Rate (CrCl) > 60 mL/min (using the Cockcroft-Gault formula):

   For women: CrCl = (140 - age) × weight (kg) × 0.85 / (72 × Scr mg/dl) For men: CrCl = (140 - age) × weight (kg) × 1.00 / (72 × Scr mg/dl)
7. Basic liver function is normal: Serum total bilirubin ≤ 1.5×ULN; AST (Aspartate Aminotransferase) ≤ 2.5×ULN; ALT (Alanine Aminotransferase) ≤ 2.5×ULN.
8. Signed written informed consent.

Exclusion Criteria:

1. Participated in another interventional clinical trial within the last 30 days;
2. Patients with severe underlying oral diseases who cannot tolerate radiation therapy;
3. Patients allergic to glutamine and thalidomide;
4. Patients receiving secondary radiation therapy to the oral area;
5. Pregnant women (confirmed by blood or urine HCG testing) or breastfeeding women, or participants of childbearing age who are unwilling or unable to take effective contraceptive measures (applicable to both male and female participants) until at least 6 months after the last trial treatment;
6. Patients with underlying peripheral neuropathy;
7. Individuals deemed by the researcher to be inappropriate for participation in this study;
8. Unwilling to participate in this study or unable to sign informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Median time for the occurrence of Grade 2 radiation-induced oral mucositis | during radiotherapy up to 4 weeks
  Median time for the occurrence of Grade 2 radiation-induced oral mucositis

SECONDARY OUTCOMES:
incidence rate of ≥grade 2 oral mucositis | during radiotherapy up to 4 weeks
  incidence rate of ≥grade 2 oral mucositis
Body mass index | during radiotherapy up to 4 weeks
  <18.5kg/m2 indicates underweight, 18.5kg/m2-23.9kg/m2 indicates normal weight, >23.9kg/m2 indicates obesity.
QOL | during radiotherapy up to 4 weeks
  Out of a total of 60 points, a score less than 20 indicates extremely poor quality of life; 21-30 points indicates poor quality of life; 31-40 points indicates average quality of life; 41-50 points indicates relatively good quality of life; 51-60 points indicates good quality of life.
adverse effects | during radiotherapy up to 4 weeks
  adverse effects

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology, Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No